CLINICAL TRIAL: NCT04576767
Title: Changes of Cognitive Function and Serum Levels of Calcium, Inflammatory Factors and Orphanin fQ in Diabetic Patients Under General Anesthesia
Brief Title: Changes of Cognitive Function and Orphanin FQ in Diabetic Patients Under General Anesthesia.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, principal investigation, Second Hospital of Shanxi Medical University
Other Study IDs: hanyi20200701
Record Dates: First submitted 2020-07-19; First posted 2020-10-06 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Cognitive Dysfunction
Keywords: The orphanin system; calcium ion; inflammatory factor
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Anesthetics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Experimental group: interventions:general anesthesia drugs:propofol、muscle relaxant、pain relievers(fentanbyl、sufentanil)
  Interventions: Other: anaesthetic
- control group: interventions:intraspinal anesthesia drugs:ropivacaine、pain relievers(fentanbyl、sufentanil)
  Interventions: Other: anaesthetic

INTERVENTIONS:
Other: anaesthetic — different states of consciousness

SUMMARY:
This study is the first to investigate the relationship between the changes of serum calcium and orphanin fq and the changes of cognitive function in patients with diabetes.To general anesthesia surgery of patients with diabetes as research group (group A), and to the non-general anesthesia surgery of diabetic patients as control group (group B), and then measured preoperative serum calcium ion concentration in patients with general anesthesia, inflammatory factor and solitary brown peptide content, intraoperative calcium ion concentration in serum, inflammatory factor and solitary brown peptide content, and postoperative serum calcium ion, inflammatory factor and solitary brown peptide content.Postoperative cognitive function were evaluated in both groups.Finally, the two groups of patients were screened and the inconsistent medical records were eliminated.Observation indicators: Endothelin, C-reactive protein, nitric oxide, interleukin-6, calcium ion concentration, orphanin fq concentration, glycated hemoglobin value and blood glucose value were observed before, during and after operation.The cognitive function of diabetic patients after surgery was observed. The cognitive function was evaluated with the cognitive function assessment scale 24 hours after surgery, respectively, and scores were obtained.Expected results: The comparison of clinical data between the control group and the study group showed that the cognitive function of patients in the study group was lower than that in the control group; the analysis showed that the serum content of orphanin fq in the study group was higher than that in the control group, the content of related inflammatory factors was higher than that in the control group, and the content of calcium ion was lower than that in the control group, and the differences were statistically significant.The results showed that when the cognitive function decreased, the content of orphanin fq increased, the corresponding inflammatory factors increased and the content of calcium decreased, indicating that the change of consciousness state and cognitive function were correlated with the orphanin fQ system.

DETAILED DESCRIPTION:
Objective: To investigate the changes of cognitive function in diabetic patients under general anesthesia, and test whether the changes of serum calcium ion, inflammatory factors and orphanin fQ are correlated. By prospective case study controlled study of diabetes (research group) general anesthesia surgery and the non-general anesthesia surgery of diabetes patients (control group), through the assessment of cognitive function and serum calcium ion, inflammation factors and the change of isolated brown peptide content to watch, in order to obtain reliable data to explore consciousness change changes of cognitive function in patients with diabetes and cognitive function in the process of the change of serum calcium ion concentration, the corresponding inflammation factors and solitary brown peptide content if there is a corresponding changes.The medical records of the patients were recorded. General information of the selected patients was recorded: gender, age, relevant medical history;Test results: blood glucose, hemoglobin , blood pressure;Drug use of patients: blood pressure drugs, hypoglycemic drugs, insulin, etc.;To observe and compare the changes of cognitive function between the control group and the study group, to detect the levels of calcium ion and orphanin fQ, and to conduct correlation analysis.To seek new theoretical basis and take corresponding treatment measures to improve the prognosis of patients with diabetic cognitive dysfunction and the quality of anesthesia surgery.

Objective: To investigate the changes of cognitive function and serum levels of calcium, inflammatory factors and orphanin fQ in diabetic patients under general anesthesia and non-general anesthesia.

Methods: the general anesthesia surgery of patients with diabetes is set to the team (group A), and to the general anesthesia surgery of diabetic patients as control group (group B), and then measured preoperative serum calcium ion concentration in patients with general anesthesia and solitary brown peptide content, intraoperative blood serum calcium ion concentration and solitary fei peptide content, and postoperative serum calcium and solitary brown peptide content. Postoperative cognitive function were evaluated in both groups.Finally, the two groups of patients were screened and the inconsistent medical records were eliminated.Observation indicators: Endothelin, C-reactive protein, nitric oxide, interleukin-6, calcium ion concentration, orphanin fq concentration, glycated hemoglobin value and blood glucose value were observed before, during and after operation.

The cognitive function of diabetic patients after surgery was observed. The cognitive function was evaluated with the cognitive function assessment scale 24 hours after surgery, respectively, and scores were obtained.

Statistical processing: Statistical Product and Service Solutions （SPSS ）21.0 statistical software was used for data analysis. Measurement data consistent with normal distribution were expressed as (mean±SD). Independent sample T-test was used for data comparison between the two groups.Repeated measurement data were compared by repeated measurement anOVA, and P < 0.05 was considered statistically significant.

Expected results: Compared with the clinical data of the control group and the study group, the cognitive function of patients in the study group was lower than that in the control group, the serum levels of orphanin fq in the analysis group were higher than those in the control group, and the levels of calcium ions in the analysis group were lower than those in the control group, and the differences were statistically significant.The results showed that when the cognitive function decreased, the content of orphanin fq increased, the content of corresponding inflammatory factors increased, and the content of calcium decreased, indicating that the change of consciousness state and cognitive function were correlated with the orphanin fQ system.

ELIGIBILITY:
Inclusion Criteria:

* The study group was diagnosed as type 2 diabetes by endocrinologist;
* Patients aged 40 or above;
* Patients with diabetes with a course of 5-10 years, 10-15 years or more;
* Duration of operation is 2-3h, American Society of Anesthesiologists (ASA)grade II-III;
* The blood glucose level of diabetic patients undergoing general anesthesia should be controlled within the normal range, and the hemoglobin of patients should be controlled within the normal range.

Exclusion Criteria:

* A definite history of central nervous system (CNS) diseases that may cause cognitive changes, such as craniocerebral trauma, craniocerebral tumor, intracranial infection, Parkinson's disease, and CNS demyelination disease;
* Mental retardation or congenital intelligence disorder, poor compliance;
* Patients with alcohol dependence, drug addiction and long-term use of mental and other drugs that affect cognitive function;
* Failure of major organs (heart, lung, liver, kidney) and critically ill patients (patients with severe trauma and infection);
* Patients with hyperthyroidism, hypothyroidism and other thyroid dysfunction and parathyroid dysfunction;
* Patients who need blood transfusion for treatment during hospitalization or have excessive blood loss during perioperative period;
* Patients with electrolyte disturbance;Patients with abnormal clotting function;
* Patients whose serum levels of endothelin, C-reactive protein, nitric oxide and interleukin-6 increased beyond the normal range after surgery.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Diabetic patients under general anesthesia, diabetic patients of different ages, diabetic patients of different course of disease, diabetic patients with different blood glucose levels
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Score of the cognitive function of diabetic patients after surgery . | change from the baseline score at 24 hours after the treatment
  The cognitive function was evaluated with the cognitive function assessment scale 24 hours after surgery, and scores were obtained.（the Montreal Cognitive Assessment, MoCA. The highest score of the test is 30 points, which is higher than or equal to 26 points is the normal level.）
the Orphanin-FQ blood level | change from the baseline Orphanin-FQ blood level at 24 hours after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guo zhen, doctor, Study Chair — Second Hospital of Shanxi Medical University
Locations (1):
- Second of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided
The consent of the participants has not been obtained